CLINICAL TRIAL: NCT05372185
Title: Expanding Reach of Evidence-based Psychotherapy for Rural Veterans With Co-occurring Anxiety and Substance Use Disorders.
Brief Title: Expanding Reach of Evidence-based Psychotherapy for Veterans With Co-occurring Anxiety and Substance Use Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Anthony H Ecker, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-48017
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Anxiety Disorders; Substance Use Disorders
MeSH Terms: conditions — Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA CALM-S (Experimental): Active psychotherapy using VA CALM-S, a weekly (9-12 sessions) cognitive behavioral therapy addressing co-occurring anxiety and substance use disorders, using disorder specific and transdiagnostic tools.
  Interventions: Behavioral: VA Coordinated Anxiety Learning and Management- Substance Use Version
- Usual Care (Active Comparator): Participants in usual care will engage with VA healthcare using standard procedures of their facility.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: VA Coordinated Anxiety Learning and Management- Substance Use Version — VA Coordinated Anxiety Learning and Management- Substance Use Version (VA CALM-S) is a cognitive behavior therapy (CBT) program that employs computer assistance to empower providers to deliver CBT with high fidelity. The computer program guides both providers and patients in a course of CBT, and in this study the content will focus on using transdiagnostic treatment elements to address co-occurring anxiety and substance use disorders.
  Arms: VA CALM-S
Behavioral: Usual care — Veterans will engage in VA care using the standard procedures of their facility.
  Arms: Usual Care

SUMMARY:
The current study seeks to better understand how to improve access to evidence-based psychotherapy (EBP) for rural Veterans with co-occurring anxiety and substance use disorders (SUD) using a web-based cognitive behavioral therapy tool (VA Coordinated Anxiety Learning and Management, Substance Use Version; VA CALM-S).

ELIGIBILITY:
Inclusion Criteria:

* current anxiety disorder diagnosis
* current SUD

Exclusion Criteria:

* current substance withdrawal such that medically supervised detoxification is necessary (determined by evaluation of substance use history and report of current symptoms),
* acute suicidality
* current delusions/hallucinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 | 12 weeks
  Self report measure of anxiety symptoms (score range 0-21), higher scores indicate greater anxiety (i.e., poorer outcome).

SECONDARY OUTCOMES:
Substance use frequency | 12 weeks
  Number of substance use days

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E DeBakey VAMC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No